CLINICAL TRIAL: NCT07350122
Title: Effect of BIS-Guided Sedation on Clinical Outcomes in Postoperative Cardiac Surgery ICU Patients: A Prospective, Randomized Controlled Trial
Brief Title: BIS in ICU Interventional Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1579
Record Dates: First submitted 2025-12-04; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgical Procedures (Postoperative Population); Critical Illness; Postoperative Complications (Cardiopulmonary); Delirium - Postoperative; Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Critical Illness; Postoperative Complications; Emergence Delirium; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-masked. Treating staff (care providers) are unblinded; outcome assessors (and data analysts) are blinded to group assignment. Participants are not specifically masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS-Guided Sedation (Experimental): Continuous BIS monitoring is visible to the care team. Sedation is titrated using BIS values plus routine clinical assessment, with instruction to avoid sustained BIS < 50.
  Interventions: Other: Device-guided sedation
- Standard Sedation with Blinded BIS (Active Comparator): Sedation is managed per standard clinical practice using validated clinical scales (e.g., RASS). BIS monitoring is performed but hidden from caregivers (not used for clinical decisions).
  Interventions: Other: standard sedation practice

INTERVENTIONS:
Other: Device-guided sedation — in addition to standard clinical sedation management, BIS monitoring will be applied in order to avoid unintended deep sedation
  Arms: BIS-Guided Sedation
Other: standard sedation practice — sedation due to standard clinical practice, using sedation scores such as RASS-Score
  Arms: Standard Sedation with Blinded BIS

SUMMARY:
This study will test whether using a Bispectral Index (BIS) monitor to guide sedation can reduce the amount of sedative medication given to adults in the intensive care unit (ICU) after cardiac surgery. BIS is a non-invasive, EEG-based monitor that shows a number from 0-100 to reflect level of consciousness. Researchers will compare BIS-guided sedation to standard sedation guided by clinical scales (such as the Richmond Agitation-Sedation Scale, RASS).

About 144 participants will be randomly assigned (1:1) to one of two groups at two hospitals in Austria (Medical University of Graz and Klinikum Wels-Grieskirchen). In the BIS group, clinicians will use BIS values and standard care to titrate sedation and will aim to avoid sustained BIS values below 50. In the control group, sedation will follow standard practices using clinical scales; BIS will be recorded but hidden from caregivers. The trial is open-label for treating staff; outcome assessors and data analysts will be blinded.

Participants will be in the study during their ICU sedation and mechanical ventilation period (typically more than 6 hours), with follow-up through ICU and hospital discharge. The primary outcome is the time-averaged dose of propofol (mg/kg/h) given during continuous ICU sedation until weaning (up to 72 hours). Secondary outcomes include duration of ventilation and sedation, depth of sedation measures, sedative and catecholamine doses, pulmonary infections (including ventilator-associated pneumonia), ICU and hospital length of stay, delirium, and in-hospital mortality.

Risks are minimal and may include mild skin irritation from forehead electrodes. Possible benefits include improved sedation management; benefits are not guaranteed. Taking part is voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing cardiac surgery with subsequent admission to the intensive care unit (e.g., valve surgery, coronary artery bypass grafting, aortic surgery)
* Planned or expected duration of invasive mechanical ventilation > 6 hours postoperatively
* Requirement for continuous sedation during ICU stay

Exclusion Criteria:

* Pre-existing neurological disorders affecting consciousness or sedation assessment (e.g., severe dementia, epileptic encephalopathy).
* Acute neurological events in the perioperative period (e.g., stroke, intracranial hemorrhage).
* Severe hepatic dysfunction (Child-Pugh Class C).
* Participation in another interventional study potentially affecting sedation or cognitive outcomes.
* Pregnancy or lactation.
* Do-not-intubate (DNI)/Do-not-resuscitate (DNR) orders or documented limitation of therapy.
* Patients in whom short-term survival is deemed unlikely due to the clinical course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
time-averaged Propofol dose during continuous ICU sedation | immediately after discontinuation of propofol
  mean Propofol infusion rate in mg/kg/h averaged over the continuous sedation period until discontinuation of Propofol (or switch to other sedative, return to OR or death)

SECONDARY OUTCOMES:
Duration of invasive mechanical ventilation | immediately after extubation
  Duration of invasive mechanical ventilation in hours
Duration of continuous sedation | immediately after extubation
  Duration of continuous sedation in hours
Incidence of pulmonary infections | at ICU discharge
  pneumonie, tracheobronchial infections
Proportion of time spent in deep sedation | immediately after discontinuation of Propofol
  Proportion of time during sedation with BIS values <50
BIS values over time | immediately after discontinuation of Propofol
  Bispectral Index (BIS) is a monitoring system providing values from 0 to 100, reflecting brain activity with 100 being fully awake an 0 indicating no brain activity (isoelectric EEG). A range of 40-60 typicallysignifies adequate general anesthesia during surgery.
Length of ICU stay | at ICU discharge
  Length of ICU stay in days
Total hospital length of stay | at hospital discharge
  Total hospital length of stay in days
In-hospital mortality | at ICU discharge
Incidence of ICU delirium | immediately after extubation
  Incidence of ICU delirium (assessed using CAM-ICU or ICDSC)
Time-averaged catecholamine dose administered (in mcg/kg/min) during continuous sedation | immediately after discontinuation of Propofol

IPD SHARING:
Plan to Share IPD: Yes
Types of data: De-identified individual participant data (IPD) underlying the primary and secondary outcomes (e.g., demographics, baseline characteristics, BIS values, sedation dosing, ventilation duration, ICU/hospital length of stay, delirium measures, adverse events).
  Supporting documents: Study protocol, statistical analysis plan (SAP), data dictionary/metadata, and analytic code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 12 months after publication of the primary results and for a period of 5 years thereafter
Access Criteria: Available to qualified researchers with a methodologically sound proposal. Requests will be reviewed by the Principal investigator. Approved requestors must:
  Sign a data use agreement (DUA) prohibiting re-identification and onward sharing.
  Obtain local IRB/ethics approval (or exemption) for the proposed analysis. Use data solely for the approved purpose and comply with GDPR and applicable data protection laws.
  Mode of access: Controlled access via the University Hospital Graz secure institutional repository. Instructions for requesting access will be provided via the study contact email: [selina.sartori@medunigraz.at]